CLINICAL TRIAL: NCT07192822
Title: Using Immersive Virtual Reality to Reduce Brief Pain During Thermal Heat Stimuli
Brief Title: Magic Bowl Virtual Reality Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Research Scientist, Human Photonics Lab, Dept of Mechanical Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VRAnalgesia2026
Record Dates: First submitted 2025-09-03; First posted 2025-09-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pain Acute
Keywords: virtual reality analgesia; pain; distraction; attention
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- One thermal stimulus (Active Comparator): participants receives a single brief thermal stimulus
  Interventions: Behavioral: One brief pain stimulus
- two thermal stimuli (Experimental): participant receives two brief thermal stimuli at the same time
  Interventions: Behavioral: Two simultaneous brief thermal stimuli
- immersive virtual reality (Active Comparator): participant receives a brief thermal stimulus while in virtual reality
  Interventions: Behavioral: Virtual Reality distraction
- No VR (Sham Comparator): brief thermal stimulus during no VR
  Interventions: Behavioral: No Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality distraction — Participants goes into an immersive virtual reality during a brief painful stimulus
  Arms: immersive virtual reality
Behavioral: No Virtual Reality — Participant receives a brief thermal stimulus during no treatment
  Arms: No VR
Behavioral: One brief pain stimulus — patient receives one brief pain stimulus with no simultaneous second stimulus
  Arms: One thermal stimulus
Behavioral: Two simultaneous brief thermal stimuli — Participants receive two brief thermal stimuli at the same time
  Arms: two thermal stimuli

SUMMARY:
Participants will rate how much pain they experience during several brief thermal stimulations at painful but tolerable temperatures participants pre-approve. During some of the stimuli participants will be in virtual reality, and during some stimuli participants will not be in VR. Sometimes participants will receive two brief stimuli at the same time.

DETAILED DESCRIPTION:
During VR, participants will put their cyberhand into a bowl of animated water and will place virtual objects in the bowl and stir the virtual water. Participants will also receive several brief thermal heat stimulations at a temperature of their choice (sometimes one stimulus, sometimes two simultaneous stimuli). During some of the stimuli participants will be in virtual reality, and some stimuli will not be in VR.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older

Exclusion Criteria:

* People how have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.
* Not enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
worst pain during one stimulus vs during two simultaneous stimuli | measured immediately after each pain stimulus
  graphic rating scale of worst pain intensity measured after one brief thermal pain stimuli, minimum = 0, maximum = 10, and measured again after two simultaenous thermal pain stimuli. In both cases, higher scores mean worse outcome

SECONDARY OUTCOMES:
worst pain during No VR vs worst pain during Virtual Reality | measured immediately after each pain stimulus
  graphic rating scale of worst pain intensity measured after one brief thermal pain stimulus with no VR, minimum = 0, maximum = 10, and measured again after one thermal pain stimuli during virtual reality. In both cases, higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: HUNTER HOFFMAN, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified aggregated summary statistics will be provided by the principle investigator upon reasonable request
Time Frame: beginning when the paper is published until Jan 1, 2030
Access Criteria: Access will be granted upon reasonable request. The requester will be emailed de-identified aggregated summary statistics provided by hunthoff9@gmail.com upon reasonable request
URL: http://www.vrpain.com

REFERENCES:
- [Background] Al-Ghamdi NA, Meyer WJ 3rd, Atzori B, Alhalabi W, Seibel CC, Ullman D, Hoffman HG. Virtual Reality Analgesia With Interactive Eye Tracking During Brief Thermal Pain Stimuli: A Randomized Controlled Trial (Crossover Design). Front Hum Neurosci. 2020 Jan 23;13:467. doi: 10.3389/fnhum.2019.00467. eCollection 2019. PMID 32038200